CLINICAL TRIAL: NCT01638611
Title: A Randomized, Double-blind, Third Party (Sponsor) Open, Placebo-controlled Study of the Tolerability and Pharmacokinetics of Single Ascending Subcutaneous Doses of HIP2B in Healthy Male Subjects
Brief Title: A Study of Subcutaneous Doses of HIP2B in Healthy Male Subjects
Acronym: HIP2B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CureDM (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TDU11656
Record Dates: First submitted 2012-07-03; First posted 2012-07-12 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Healthy male volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIP2B (Active Comparator): Six subjects per dosing cohort will receive HIP2B
  Interventions: Drug: HIP2B
- Placebo (Placebo Comparator): Two subjects per dosing cohort will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HIP2B — Total daily doses of 60, 120, 240, 480, and 720 mg are planned in five separate dosing cohorts. Single or split dose (depending on dose volume) will be given by subcutaneous injection in the abdomen to six subjects per dosing cohort.
  Arms: HIP2B
Drug: Placebo — Equal volumes of placebo will be given by subcutaneous injection in the abdomen to 2 randomized subjects per dosing cohort.
  Arms: Placebo

SUMMARY:
HIP2B is the stabilized form of the Human proIslet Peptide (HIP). Human proIslet Peptide is the human homolog of Islet Neogenesis Associated Protein (INGAP) peptide, which has shown signals of efficacy in type 1 and type 2 diabetes mellitus. In a mouse model of diabetes, repeat dose treatment with HIP results in new islet formation and improvement in blood glucose measurements.

HIP2B is being developed for the treatment of type 1 and type 2 diabetes mellitus.

The present clinical trial protocol proposes the first administration of HIP2B to humans with the goal of exploring the tolerability, safety and PK of HIP2B following subcutaneous single ascending doses.

DETAILED DESCRIPTION:
Primary Outcome:

To assess the tolerability and safety after subcutaneous single ascending doses of HIP2B in healthy male subjects. Adverse events including local injection site reactions/pain will be assessed during the study. Ongoing adverse events will be followed to resolution or for 30 days (whichever is sooner). Clinical laboratory evaluations including amylase and lipase will be reviewed. Vital signs and ECGs will be used to evaluate subject safety.

Secondary Outcome:

To assess the pharmacokinetics (including Cmax, AUClast, AUC0-∞, tmax, t1/2, tlag) in healthy male subjects after subcutaneous single ascending doses of HIP2B.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy, male, between 19 and 45 years inclusive.
* Subject's body weight is between 50.0 and 100.0 kg inclusive and body mass index (BMI) is between 18.0 and 31.6 kg/m2 inclusive.
* Subject is certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination) by the study doctor.
* Subject has normal vital signs after 10 minutes resting in supine position:

  * 95 mmHg ≤ systolic blood pressure ≤ 140 mmHg
  * 45 mmHg ≤ diastolic blood pressure ≤ 90 mmHg
  * 40 beats per minute ≤ heart rate ≤100 beats per minute
* Subject has a normal standard 12-lead ECG after 10 minutes resting in supine position; 120 ms < PR < 220 ms, QRS < 120 ms, QTc ≤ 450 ms. Subject must be fasting.
* Laboratory parameters for the subject are within the normal range (or defined screening threshold for the Investigative site), unless the Investigator considers an abnormality to be not clinically significant for healthy subjects; however serum creatinine, alkaline phosphatase, hepatic enzymes (AST/ ALT, amylase, lipase, and fractional bilirubin (direct and indirect) should not exceed the upper laboratory norm).
* Male subjects must continue to use their approved contraceptive method and to refrain from donating semen for 30 days after participating in the study.
* The subject has given written informed consent prior to any study related procedures being performed.
* The subject is not under any administrative or legal supervision.

Exclusion Criteria:

* The subject has any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteo-muscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* The subject has frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* The subject has significant blood loss or blood donation, within 56 days prior to IP administration.
* The subject exhibits symptomatic hypotension, whatever the decrease in blood pressure, or asymptomatic postural hypotension defined by a decrease in systolic blood pressure ≥ 20 mmHg within 3 minutes when changing from the supine to the standing position.
* The subject has the presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* The subject has a history or presence of drug or alcohol abuse (alcohol consumption > 2 drinks per day).
* The subject smokes more than 5 cigarettes or equivalent per day, unable to stop smoking during the days the subject is confined or returning for study related testing.
* Excessive consumption of beverages with xanthine bases (> 4 8 ounce glasses per day) including energy drinks, weight loss drinks, protein mixes (i.e. for body building), etc.
* Any medication, herbal supplement or other natural products (including St John's Wort) within 14 days before the Day 1 visit or within 5 times the elimination half-life or pharmacodynamic half-life of that drug, whichever is longest; any vaccination within the last 28 days. This includes taking analgesics 2 days before Day 1 visit which will interfere with pain assessment.
* Any subject who, in the judgment of the Investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any subject participating in another clinical trial of an investigational therapy (including placebo) within 30 days of screening or 5 half-lives of the study medication, whichever is longer.
* Any subject who cannot be contacted in case of emergency.
* Any subject who is the Investigator or any Sub-Investigator, Research Assistant, Pharmacist, Study Coordinator, or other staff thereof, directly involved in the conduct of the protocol.
* Any subject with a history or presence of any skin condition that would interfere with injection site assessments (including tattoos) and no umbilical piercings.
* Positive results on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive urine ethanol test.
* Any subject with either amylase or lipase levels above the upper laboratory norm
* Any subject with previous history of pancreatitis or known gallbladder disease (including gallstones and gallstone attacks; gallbladder removal will not exclude subject from participating).
* Any subject with prior exposure to INGAP peptide

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability and safety after subcutaneous single ascending doses of HIP2B. | Each dosing cohort will have a study duration of 7 days (±2 days). PK data will be reviewed 11 days after dosing.
  The dose escalation will be guided by safety and tolerability (includes AEs, medical assessments, clinical lab evaluation, and PK). Starting with a dose of 60 mg, a decision to proceed to the next higher "n+1" dose will be made jointly by the Medical Monitor, Sponsor and the Investigator based on blinded safety and tolerability data up to at least 24 hours post dose (Day 2) of at least 6 out of 8 subjects of dose level cohort "n".

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No